CLINICAL TRIAL: NCT00399152
Title: An Open-Label Phase I Study of the Safety of Perifosine in Combination With Sunitinib Malate for Patients With Advanced Cancers
Brief Title: Perifosine + Sunitinib Malate for Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 125
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2011-11

CONDITIONS: Renal Cancer; GIST
Keywords: Perifosine; Sunitinib Malate; Renal cancer; GIST; advanced cancers
MeSH Terms: conditions — Kidney Neoplasms | interventions — perifosine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perifosine+Sunitinib malate (Experimental)
  Interventions: Drug: Perifosine; Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Perifosine — Perifosine Oral Dose
Drug: Sunitinib Malate — Sunitinib oral dose

SUMMARY:
This study is a Phase I trial in two parts. In part 1, a MTD to the combination of perifosine and sunitinib malate will be determined. In part 2, with the MTD as a starting point, a group of patients will be accrued with the goal of ensuring that they will be able to tolerate at least two courses of therapy, which would make them evaluable for response in a Phase II study.

DETAILED DESCRIPTION:
This study is a Phase I trial in two parts. In part 1, an MTD to the combination of perifosine and sunitinib malate will be determined. In some previous trials with perifosine and other biologic agents, doses determined in Phase I studies are not as well tolerated in larger groups of patients when response is an endpoint. Thus in part 2, with the MTD as a starting point, a group of patients will be accrued with the goal of ensuring that they will be able to tolerate at least two courses of therapy, which would make them evaluable for response in a Phase II study. As a secondary endpoint, the effects of the combination of perifosine and sunitinib malate will be evaluated for response rate and time to progression. The pharmacokinetics of the combination of the study drugs will be measured.

For the purposes of this study, one cycle of therapy will be defined as 6 weeks. Patients will take one 50 mg tablet of perifosine one to three times a day and sunitinib malate once a day for 4 out of 6 weeks. Patients may need anti-emetics and/or anti-diarrheals. Patients will be evaluated for progression or response at 12-week intervals.

Patients who experience toxicity may continue on treatment with doses delayed or reduced.

All patients should continue therapy unless disease progression is documented on two occasions at least four weeks apart.

Part 1 of this Phase I study will accrue from six to 24 patients depending on the number of dose levels evaluated. Up to six patients will be treated at each dose level. A dose limiting toxicity (DLT) will be defined as:

* Grade 3 or greater non-hematologic toxicity
* Grade 4 hematologic toxicity

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically confirmed diagnosis of renal tumor or GIST are eligible for this protocol. Patients with other solid tumor types must have their cases reviewed by the OCOG medical monitor.
* The physician must believe that the patient's course and the growth rate of the tumor are such that the patient would feel comfortable continuing treatment for 12 weeks even if there is a transient period of modest tumor growth during the first weeks following the initiation of perifosine and sunitinib malate treatment.
* Patients must have a life expectancy of more than 6 months.
* Patients may have received prior sorafenib or sunitinib malate.
* Patients may have measurable or evaluable disease.
* Patients should have a performance status of 0 to 1 according to the ECOG criteria. However, patients with ECOG performance status of 2 may be admitted with approval from the study chairman or medical monitor.
* Patients must have adequate organ and marrow function, unless in the opinion of the treating investigator, the abnormality is related to tumor and the study chairman or medical monitor agree the abnormality is unlikely to affect the safety of perifosine and/or sunitinib use.
* Patients must have recovered from acute toxicity related to prior therapy including surgery or radiotherapy, excluding alopecia.
* Patients must be able to ingest oral medications or to obtain them through a gastrostomy tube.
* Patients must be at least 18 years of age.
* Patients must have ability to understand and the willingness to sign a written informed consent document.
* LVEF greater than or equal to 50%.

Exclusion Criteria:

* Rapidly progressing disease, as defined by progression within 8 weeks of initiation of the previous regimen
* Patients who have had more than three prior systemic therapies, including biologics, are excluded unless prior approval is obtained from the medical monitor
* Patients receiving any other investigational agents or devices
* Patients initiating a treatment for their cancer within the last two months who will be continued concomitantly with perifosine
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements
* Patients currently taking strong inhibitors of the CYP3A4 family (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole) AND inducers of the CYP3A4 family (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's Wort) because of possible pharmacokinetic interactions with sunitinib. Patients who are no longer taking strong CYP3A4 inhibitors and/or inducers are ineligible unless they have discontinued use 4 weeks prior to beginning therapy.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), or New York Heart Association class II-IV congestive heart failure
* Female patients who are pregnant or lactating are ineligible. All females of childbearing potential must have a negative serum pregnancy test within 72 hours of treatment. Men and women of childbearing potential must agree to employ adequate contraception to prevent pregnancy while on therapy and for 4 weeks after the completion of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Toxicities | every 6 weeks

REFERENCES:
- [Result] Preliminary results / Journal of Clinical Oncology, 2008 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 26, No 15S (May 20 Supplement), 2008: 14565